CLINICAL TRIAL: NCT07018466
Title: Tele-Exercise in Veterans With Military Exposure
Brief Title: Tele-Exercise for MERP
Acronym: TEMPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARA-010-24F
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Burn Pit Exposure
Keywords: Exercise; Cardiopulmonary; Military Exposure
MeSH Terms: conditions — Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Tele-exercise or standard of care control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-exercise (Active Comparator): Exercise training 3x/week at home. Sessions include circuit exercises of aerobic and resistive training stations which are led remotely.
  Interventions: Other: Tele-exercise
- Standard of Care (Placebo Comparator): Health education discussions and lectures 2-3x/week led remotely.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Tele-exercise — Exercise training 3x/week at home. Sessions include circuit exercises of aerobic and resistive training stations which are led remotely.
  Arms: Tele-exercise
Other: Standard of Care — Health education discussions and lectures 3x/week led remotely.
  Arms: Standard of Care

SUMMARY:
During Operations Desert Shield and Desert Storm, Veterans in combat were exposed to a variety of airborne hazards, including oil well fire smoke, emissions from burn pits, and other substances associated with negative health outcomes, including cardiovascular and pulmonary disease and cancer. More than 40% of Veterans enrolled in the VA's Airborne Hazards and Open Burn Pit Registry (AHOBPR) report functional limitations, such as difficulty running short distances. Veterans with burn pit exposures will benefit from physical activity interventions designed to improve functional ability and overall quality of life. Veterans with significant exposure to burn pits during their overseas military service will have a detailed documentation of their limitations and participate in either a 12-week coach-led tele-exercise intervention or standard of care. This project is designed to improve functional mobility and could be implemented for Veterans with burn pit exposure.

DETAILED DESCRIPTION:
The most ubiquitous air born hazards resulting from recent conflicts is likely emissions from burn pits used for slow disposal of a variety of wastes, including plastics, petroleum products, metal, rubber, medical waste, and human waste. Burn pits have been used as a waste disposal practice by the United States military for several decades but were more prominent and widespread in the recent conflicts in Iraq and Afghanistan. The burning of these wastes produces toxins that have been demonstrated to produce toxicity in animal and human models and to increase the risk of cardiopulmonary disease in large, population-based studies of Veterans. These include small particulate matter (PM2,5), airborne metal particles, volatile organic compounds (VOCs), and specific byproducts of burnt petroleum products, including polycyclic aromatic hydrocarbons (PAHs).

The long-term health effects of exposure to these toxins are incompletely understood, and the subject of intense research. Increased incidence of cardiopulmonary disease is a major concern in exposed Veterans, with an increased risk of systemic hypertension, COPD, and asthma, all having been recently reported based on a large analysis of Veteran records. Dyspnea is a core symptom linking the pleotropic health effects associated with airborne hazards exposure. A recent study of nearly 2,000 Veterans demonstrated associations between dyspnea and burn pit exposure and exposure to military dusts, gases, and fumes, as well as associations between burn pit exposure and chronic bronchitis.

Among participants in the large-scale Millennium Cohort Study, Veterans who had been deployed reported shortness of breath more frequently than those who were not deployed. As a result, a federally chartered multisite program, the Post-Deployment Cardiopulmonary Evaluation Network (PDCEN), was created specifically to evaluate the causes of underlying exercise intolerance and dyspnea in this group. While this program self-selects for deployed Veterans with symptoms, the magnitude of exercise intolerance in this group is marked.

The investigators hypothesize that Veterans within the VA's Airborne Hazards and Open Burn Pit Registry (AHOBPR) have poor physical function and mobility, and high levels of dyspnea and fatigue. The investigator's global hypothesis is that exercise rehabilitation will improve functional mobility and reduce dyspnea and fatigue in Veterans with military burn pit exposure.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age > or equal to 40 years
* Self-reported exposure to burn pits and/or burn pit smoke during overseas military deployment (at least 6 hours per day during one or more deployments of at least three months)
* ability to interact with study staff using video conferencing technology
* ability to provide written informed consent

Exclusion Criteria:

* Musculoskeletal or medical conditions which preclude participation in a tele-exercise program
* Active severe mental health or psychiatric issues, including suicidality
* Severe pulmonary disease (chronic supplemental oxygen), or lobectomy or greater resection
* Myocardial infarction (within 3 months), or exertional or unstable angina
* Uncontrolled systemic hypertension, defined as resting systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 at time of most recent evaluation at time of recruitment
* Active systemic treatment for cancer
* Acute care hospitalization within the last 90 days
* End-stage liver or renal disease
* Any other medical or psychiatric condition that would preclude safe participation in tele-exercise, according to the judgment of the investigators

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in VO2peak | Baseline and 12 weeks intervention or control
  physical fitness, units are ml/kg/min
Change in 6-minute walk test | Baseline and 12-weeks intervention or control
  distance, units are m

SECONDARY OUTCOMES:
Change in 2-minute step test | Baseline and 12-weeks intervention or control
  physical function, units are number of times

CONTACTS AND LOCATIONS:
Overall Officials: Alice S. Ryan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No